CLINICAL TRIAL: NCT02612480
Title: The Effect of Ticagrelor on the Inflammatory Response to Human Endotoxemia
Brief Title: Ticagrelor in Human Endotoxemia Response to Human Endotoxemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Peter Pickkers, Prof. Dr. Peter Pickkers, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: tica-lps; 2014-005537-30 (EudraCT Number); NL51923.091.14 (Other: CCMO)
Record Dates: First submitted 2015-11-03; First posted 2015-11-23 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Endotoxemia
Keywords: endotoxin; LPS; ticagrelor; clopidogrel; acetylsalicyclic acid; placebo
MeSH Terms: conditions — Endotoxemia | interventions — Ticagrelor; Clopidogrel; acetylsalicylic acid lysinate; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ticagrelor and acetylsalicylic acid (Experimental): 7 day treatment with ticagrelor 2x90mg after a loading dose of 180 mg and acetylsalicyclic acid 1x80mg after a loading dose of 160 mg.
  Interventions: Drug: ticagrelor; Drug: Acetylsalicylic acid lysinate
- Clopidogrel and acetylsalicylic acid (Active Comparator): 7 day treatment with clopidogrel x75 mg after a loading dose of 300 mg and acetylsalicyclic acid 1x80mg after a loading dose of 160 mg
  Interventions: Drug: Clopidogrel; Drug: Acetylsalicylic acid lysinate
- Placebo and acetylsalicylic acid (Placebo Comparator): 7 day treatment with placebo and acetylsalicyclic acid 1x80mg after a loading dose of 160 mg
  Interventions: Drug: Acetylsalicylic acid lysinate; Drug: Placebo
- Placebo (Placebo Comparator): 7 day treatment with 2 placebos
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ticagrelor — 7 day treatment of ticagrelor 2dd90mg after a loading dose of 180mg
  Other Names: brillique
  Arms: Ticagrelor and acetylsalicylic acid
Drug: Clopidogrel — 7 day treatment of clopidogrel 1d75mg after a loading dose of 300mg
  Other Names: Plavix
  Arms: Clopidogrel and acetylsalicylic acid
Drug: Acetylsalicylic acid lysinate — 7 day treatment of acetylsalicyclic acid 1d80mg after a loading dose of 160mg
  Other Names: Aspirin
  Arms: Clopidogrel and acetylsalicylic acid; Placebo and acetylsalicylic acid; Ticagrelor and acetylsalicylic acid
Drug: Placebo — 7 day treatment with placebo
  Arms: Placebo; Placebo and acetylsalicylic acid

SUMMARY:
Rationale:

In patients suffering a myocardial infarction the P2Y12 receptor antagonists prasugrel and ticagrelor improve outcome and prognosis compared to clopidogrel. Moreover, ticagrelor lowers mortality from pulmonary infections and sepsis, which cannot solely be explained by its platelet-inhibiting effect. An effect on the inflammatory response in the setting of acute myocardial might underlie this phenomenon and if substantiated support a novel beneficial mechanism of the new the P2Y12 receptor antagonists.

Objective:

To study whether ticagrelor, added to acetylsalicylic acid, modulates the inflammatory response to the administration of lipopolysaccharide (LPS) in humans in vivo, and to compare this effect with the P2Y12 antagonist clopidogrel.

Study design:

Prospective randomized placebo-controlled trial, according to a PROBE design (prospective randomized open blinded-endpoint study).

Study population:

Forty healthy male volunteers aged ≥ 18 and ≤ 35 years. Intervention (if applicable): Participants will be randomized to receive either placebo (twice daily), acetylsalicylic acid (80 mg once daily, after a loading dose of 160 mg) + placebo (once daily), acetylsalicylic acid (80 mg once daily, after a loading dose of 160 mg) + ticagrelor (90 mg twice daily, after a loading dose of 180 mg) or acetylsalicylic acid (80 mg once daily, after a loading dose of 160 mg)+ clopidogrel (75 mg once daily, after a loading dose of 300mg).

Main study parameters/endpoints:

Endpoints: area under the curve of the proinflammatory cytokines TNF-alpha, IL6, IL-10, IL1ra IL-8, IL-1β, MCP-1 MIP-1a, MIP-1b en IFN; peak concentrations of the various cytokines; plasma concentration of HMGP1; platelet-monocyte complex formation and markers of platelet function; plasma concentration of adenosine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 35 years
* Male
* No known current medical/psychiatric diseases

Exclusion Criteria:

* History, signs or symptoms of any cardiovascular disease
* History of chronic obstructive pulmonary disease (COPD) or asthma
* History of hemorrhagic diathesis, or any other disorder associated with increased risk of bleeding
* Previous spontaneous vagal collapse
* Use of any medication
* Smoking
* Liver enzyme abnormalities (defined as ALAT and/or ASAT > twice upper limit of normality)
* Thrombocytopenia (<150*109

  /ml) or anemia (haemoglobin < 8.0 mmol/L)
* Any obvious disease associated with immune deficiency
* Febrile illness in the week before the LPS challenge
* Hypersensitivity to ticagrelor or any excipients
* Active pathological bleeding
* History of intracranial haemorrhage
* History of dyspepsia
* quantitative bleeding assessment tool (BAT) score >3 (see Appendix 1)
* Participation in another drug trial or donation of blood 3 months prior, until 3 months after the planned LPS challenge
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block, third degree atrioventricular block or a complex bundle branch block
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90)
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50)
* Renal impairment (defined as MDRD < 60 ml/min)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
concentration plasma TNFalpha (pg/ml) | measured after challenge with endotoxin at day 7 of medication
  measured with Luminex assay

SECONDARY OUTCOMES:
concentration plasma IL-6 (pg/ml) | measured after challenge with endotoxin at day 7 of medication
  measured with Luminex assay
concentration plasma IL-8 (pg/ml) | measured after challenge with endotoxin at day 7 of medication
  measured with Luminex assay
concentration plasma IL-10 (pg/ml) | measured after challenge with endotoxin at day 7 of medication
  measured with Luminex assay
concentration plasma IL-1RA (pg/ml) | measured after challenge with endotoxin at day 7 of medication
  measured with Luminex assay
concentration plasma IL-1beta (pg/ml) | measured after challenge with endotoxin at day 7 of medication
  measured with Luminex assay
concentration plasma MCP-1(pg/ml) | measured after challenge with endotoxin at day 7 of medication
  measured with Luminex assay
concentration plasma MIP-1a(pg/ml) | measured after challenge with endotoxin at day 7 of medication
  measured with Luminex assay
concentration plasma MIP-1b(pg/ml) | measured after challenge with endotoxin at day 7 of medication
concentration plasma IFNgamma(pg/ml) | measured after challenge with endotoxin at day 7 of medication
  measured with Luminex assay
plasma adenosine | measured after challenge with endotoxin at day 7 of medication
platelet monocyte complexes | measured after challenge with endotoxin at day 7 of medication
  flowcytometric determination of monocytic load with platelets
platelet neutrophil complexes | measured after challenge with endotoxin at day 7 of medication
  flowcytometric determination of neutrophil load with platelets
platelet reactivity | measured after challenge with endotoxin at day 7 of medication
  ex vivo stimulation of platelets with ADP and collagen, response measured as P-selectin and fibrinogen)
monocytic tissue factor expression | measured after challenge with endotoxin at day 7 of medication
  tissue factor expression on monocytes as measured by flow cytometry
monocytic HLA-DR expression | measured after challenge with endotoxin at day 7 of medication
  as measured by flow cytometry
CD14/16 ratio | measured after challenge with endotoxin at day 7 of medication
  measured with flow cytometry
platelet von Willebrandfactor expression | measured after challenge with endotoxin at day 7 of medication
  measured with flow cytometry
VASP-P | difference between measurement prior to start of study drug after challenge with endotoxin at day 7 of medication
  ELISA
symptoms during endotoxin day | measured after challenge with endotoxin at day 7 of medication
  6 point likert scale
blood pressure | measured after challenge with endotoxin at day 7 of medication
  mmHg
temperature | measured after challenge with endotoxin at day 7 of medication
  tympanic temperature

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center; Niels Riksen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Intensive Care Medicine, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands